CLINICAL TRIAL: NCT01843556
Title: A Phase 1 Study of E2022 Tape Formulation for Different Application Sites and Intervals
Brief Title: A Phase 1 Study of E2022 Tape Formulation for Different Application Sites and Intervals in Japanese Healthy Elderly Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2022-J081-003
Record Dates: First submitted 2013-04-25; First posted 2013-04-30 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2014-02

CONDITIONS: Healthy Elderly Male
MeSH Terms: interventions — Donepezil

ARMS (1):
- E2022 Tape Formulation (Experimental)
  Interventions: Drug: E2022 Tape Formulation

INTERVENTIONS:
Drug: E2022 Tape Formulation — E2022 tape formulation applied to different application sites and at different intervals in Japanese healthy elderly males
  Other Names: Donepezil

SUMMARY:
A phase 1 study of E2022 tape formulation in healthy elderly males to evaluate the safety and pharmacokinetics.

ELIGIBILITY:
Inclusion criteria:

1. Male non-smokers (not smoking at least 4 weeks before Period 1) aged 65 years or older at informed consent
2. BMI at screening is 18.5 kg/m2 or above - below 28.0 kg/m2
3. Written informed consent
4. Given full explanation of this study and is willing to and able to comply with the protocol requirements

Exclusion criteria:

1. Have a current or past history of disorder requiring medical treatment within 8 weeks before the first application or infection within 4 weeks before the first application
2. Have a disorder within 4 weeks before the first application which affects the evaluation of study drug such as psychiatric, gastrointestinal, hepatic, renal, respiratory, endocrinological, hematological, neurological or cardiovascular system, or congenital metabolic abnormality
3. Have a history of gastrointestinal surgery (e.g., liver, kidney, digestive tract) which affects the pharmacokinetics of study drug,
4. Have a history of treatment-requiring drug or food allergy or seasonal allergy at screening
5. Had caffeine-containing food or drink or alcohol within 72 hours before study drug application in Period I
6. Had nutritional supplements, herbal preparations (including oriental medicines) or others (e.g., grapefruit-containing food or beverage) which may affect drug metabolizing enzymes and transporters, within 1 weeks before Period I
7. Have used liquid products (including cosmetics) on study application sites (back, upper limb, chest), patch, tape or bandage, within 4 weeks before Period 1
8. Present or past clinical signs of skin hypersensitivity to topical product or atopic dermatitis
9. Excessively hairy or have shaved at application sites (back, upper limb, chest) within 4 weeks before Period 1
10. Eczema, dermatitis, abnormal pigmentation, injury, or scar at application sites which may affect the evaluation of skin symptoms

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events | 168 hours after the end of application

SECONDARY OUTCOMES:
Maximal Drug Concentration (CMax) | 216 hours after the end of application
Area Under the Plasma Concentration-Time Curve (AUC) | 216 hours after the end of application
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 216 hours after the end of application
Plasma Decay Half-Life (t1/2) | 216 hours after the end of application

CONTACTS AND LOCATIONS:
Overall Officials: Hidetaka Hiramatsu, Study Director — Eisai Co., Ltd.
Locations (1):
- Kagoshima, Japan